CLINICAL TRIAL: NCT00910962
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety of 12 Weeks of Dosing With GW856553 and Its Effects on Inflammatory Markers, Infarct Size, and Cardiac Function in Subjects With Myocardial Infarction Without ST-segment Elevation
Brief Title: A Study to Evaluate the Safety of 12 Weeks of Dosing With GW856553 and Its Effects on Inflammatory Markers, Infarct Size, and Cardiac Function in Subjects With Myocardial Infarction Without ST-segment Elevation
Acronym: Solstice
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 111810
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Results first posted 2017-10-27 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-09

CONDITIONS: Acute Coronary Syndrome
Keywords: NSTEMI, acute coronary syndrome, p38 MAPK inhibitor, GW856553, percutaneous coronary intervention
MeSH Terms: conditions — Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment A (Experimental): 7.5 mg GW856553 starting dose, followed 12 hours later by 7.5mg twice daily for 12 weeks
  Interventions: Drug: GW856553
- Treatment B (Experimental): 15 mg GW856553 starting dose, followed 12 hours later by 7.5mg twice daily for 12 weeks
  Interventions: Drug: GW856553
- Treatment C (Placebo Comparator): Placebo twice daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GW856553 — 7.5 mg GW856553 starting dose, followed 12 hours later by 7.5mg BID
  Arms: Treatment A
Drug: GW856553 — 15 mg GW856553 starting dose, followed 12 hours later by 7.5mg BID
  Arms: Treatment B
Drug: Placebo — Placebo
  Arms: Treatment C

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel group, multi-center study to evaluate initial safety and efficacy of GW856553 in subjects with NSTEMI. Up to approximately 525 subjects will be randomized to meet the MRI recruitment target (90 subjects in substudy.) All subjects will continue to receive the local standard of care for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a NSTEMI, defined as: symptoms (e.g. chest pain, dyspnea) consistent with acute coronary syndrome, lasting at least 10 minutes, with most recent symptoms occurring within the 24 hours prior to presentation, without persistent ST-segment elevation on admission 12-lead ECG, and with Troponin (T or I) above the upper limit of normal (ULN) for the local institution within 18 hours of presentation.
* Subject able to be randomized within 18 hours of presentation.
* Subjects to be managed with an early invasive strategy, with PCI likely to occur at least 2 hours after the start of dosing [subjects who do not undergo PCI will not be withdrawn from the study].
* Male or female subject who is 45 years of age or older.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) greater than 40 MlU/ml and estradiol less than 40 pg/ml (less than 140 pmol/L) is confirmatory), or child-bearing potential and agrees to use one of the contraception methods listed in the protocol for the duration of dosing and until the first follow-up visit (approximately 2 weeks post last-dose).
* Negative urine or serum pregnancy test (in women of child-bearing potential only).
* Male subjects must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until the first follow-up visit (approximately 2 weeks post last-dose).
* QTcB or QTcF greater than 530 msec.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* History of severe heart failure defined as NYHA class III or IV or those with known severe LV dysfunction [ejection fraction less than 30%] regardless of symptomatic status.
* Suspected aortic dissection.
* Severe aortic stenosis or other severe valvular disease.
* Current known life-threatening condition other than vascular disease (e.g. severe chronic airways disease) that may prevent a subject from completing the study.
* Subjects with rheumatoid arthritis, connective tissue disorders and other conditions known to be associated with active chronic or acute inflammation (e.g. inflammatory bowel disease, osteomyelitis, pneumonia, etc.). Intermittent conditions treated with short-term oral antibiotics (e.g. typical URI) or conditions that are not currently exacerbated (e.g. gout with no current flair) may be included.
* History of myopathy or rhabdomyolysis.
* Current or chronic history of liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Known to be Hepatitis B or Hepatitis C positive.
* Current or anticipated use of systemic steroids (oral or IV). Inhaled, intranasal and topical steroids are allowed. A single prophylactic dose of systemic steroid is allowed at time of PCI for subjects with contrast allergy.
* Current or anticipated use of BCRP substrates with a narrow therapeutic index (e.g. daunorubicin, doxorubicin, topotecan, mitoxantrone).
* Previously diagnosed cancer that has not been in complete remission for at least 5 years. Localized carcinomas of the skin and carcinoma in situ of the cervix that have been resected or ablated for cure are not exclusionary..
* Known alcohol or drug abuse within the past 6 months.
* Previous exposure to GW856553.
* Use of another investigational product within 30 days or 5 half-lives (whichever is the longer) preceding the first dose of IP in the current study.
* Any other subject whom the Investigator deems unsuitable for the study (e.g., due to either medical reasons, laboratory abnormalities, expected study medication non-compliance).
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Previous MI or coronary artery bypass graft (CABG) surgery.
* History of kidney transplant or a history of contrast nephropathy.
* Contraindication to MRI scanning (as assessed by local MRI safety questionnaire) which includes but is not limited to: intracranial aneurysm clips or other metallic objects; history of intra-orbital metal fragments that have not been removed by an MD; pacemakers and non-MR compatible heart valves; inner ear implants; history of claustrophobia in MR.
* Allergy to MRI contrast enhancement agent (gadolinium).
* Estimated creatinine clearance by Cockcroft-Gault formula < 30 mL/min.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2009-10-08 (Actual); Primary Completion 2012-03-06 (Actual); Study Completion 2012-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (97):
- United States (30):
  - GSK Investigational Site, Anchorage, Alaska
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Elyria, Ohio
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Camp Hill, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Oak Ridge, Tennessee
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Round Rock, Texas
  - GSK Investigational Site, Victoria, Texas
- Australia (8):
  - GSK Investigational Site, Kogarah, New South Wales
  - GSK Investigational Site, Liverpool, New South Wales
  - GSK Investigational Site, Brisbane, Queensland
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Woodville South, South Australia
  - GSK Investigational Site, Launceston, Tasmania
  - GSK Investigational Site, Fremantle, Western Australia
  - GSK Investigational Site, Perth, Western Australia
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Terrebonne, Quebec
- Germany (32):
  - GSK Investigational Site, Bad Krozingen, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Rastatt, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Bad Nauheim, Hesse
  - GSK Investigational Site, Darmstadt, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Limburg an der Lahn, Hesse
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Oldenburg, Lower Saxony
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Bielefeld, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Leverkusen, North Rhine-Westphalia
  - GSK Investigational Site, Neuss, North Rhine-Westphalia
  - GSK Investigational Site, Wuppertal, North Rhine-Westphalia
  - GSK Investigational Site, Worms, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Pirna, Saxony
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Bad Berka, Thuringia
  - GSK Investigational Site, Erfurt, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- India (4):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Calicut
  - GSK Investigational Site, Pune
- Netherlands (4):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Arnhem
  - GSK Investigational Site, Nieuwegein
  - GSK Investigational Site, Tilburg
- Poland (3):
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Radom
  - GSK Investigational Site, Warsaw
- Spain (5):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Jerez (Cadiz)
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Santiago de Compostela
- United Kingdom (7):
  - GSK Investigational Site, Brighton, East Sussex
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Clydebank
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, London
  - GSK Investigational Site, Paddington, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Newby LK, Marber MS, Melloni C, Sarov-Blat L, Aberle LH, Aylward PE, Cai G, de Winter RJ, Hamm CW, Heitner JF, Kim R, Lerman A, Patel MR, Tanguay JF, Lepore JJ, Al-Khalidi HR, Sprecher DL, Granger CB; SOLSTICE Investigators. Losmapimod, a novel p38 mitogen-activated protein kinase inhibitor, in non-ST-segment elevation myocardial infarction: a randomised phase 2 trial. Lancet. 2014 Sep 27;384(9949):1187-95. doi: 10.1016/S0140-6736(14)60417-7. Epub 2014 Jun 12. PMID 24930728
- [Derived] Melloni C, Sprecher DL, Sarov-Blat L, Patel MR, Heitner JF, Hamm CW, Aylward P, Tanguay JF, DeWinter RJ, Marber MS, Lerman A, Hasselblad V, Granger CB, Newby LK. The study of LoSmapimod treatment on inflammation and InfarCtSizE (SOLSTICE): design and rationale. Am Heart J. 2012 Nov;164(5):646-653.e3. doi: 10.1016/j.ahj.2012.07.030. Epub 2012 Oct 16. PMID 23137494
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 111810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 535 participants, with myocardial infarction without ST segment elevation, were randomized to the study of which 526 participants received at least one dose of study drug. The study was conducted at 83 centers, from 08 October 2009 to 06 March 2012.
Groups:
- Placebo (P): Eligible participants received matching placebo, orally twice daily for 12 weeks.
- Losmapimod 7.5 mg (A): Eligible participants received oral losmapimod 7.5 milligrams (mg) starting dose, followed 12+/-4 hours, later by losmapimod 7.5 mg twice daily maintenance dose for 12 weeks (referred to as non-loading dose group).
- Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B): Eligible participants received oral losmapimod 15 mg starting dose, followed 12+/-4 hours, later by losmapimod 7.5 mg twice daily maintenance dose for 12 weeks (referred to as loading dose group).
Period: Overall Study
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B)
Started | 135 | 199 | 192
Completed | 92 | 121 | 116
Not Completed | 43 | 78 | 76
Not completed — Adverse Event | 5 | 20 | 17
Not completed — Protocol Violation | 1 | 3 | 3
Not completed — Lost to Follow-up | 0 | 3 | 1
Not completed — Physician Decision | 0 | 6 | 6
Not completed — Withdrawal by Subject | 25 | 32 | 32
Not completed — Reached defined stopping criteria | 12 | 14 | 17

BASELINE CHARACTERISTICS:
Population: The race of one participant each in treatment A and treatment B were unknown.
Groups:
- Losmapimod 7.5 mg (A): Eligible participants received oral losmapimod 7.5 mg starting dose, followed 12+/-4 hours, later by losmapimod 7.5 mg twice daily maintenance dose for 12 weeks (referred to as non-loading dose group).
- Total: Total of all reporting groups
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | Total
Number analyzed (Participants) | 135 | 199 | 192 | 526
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.4 (10.29) | 62.6 (11.03) | 64.6 (10.50) | 63.5 (10.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 52 | 57 | 149
  Male | 95 | 147 | 135 | 377
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 0 | 3
  Asian | 4 | 4 | 9 | 17
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3 | 6
  Black or African American | 2 | 6 | 5 | 13
  White | 128 | 183 | 174 | 485
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE was any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE was any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment.
Time Frame: Up to Week 14
Population: Safety Population consisted of all participants randomized to treatment, who had taken at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- A and B Combined (C): A combined data for eligible participants from arm A and arm B were presented.
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 135 | 199 | 192 | 391
Participants
  Any AE | 97 | 138 | 131 | 269
  Any SAE | 32 | 51 | 43 | 94

2. Primary Outcome: Number of Participants With Any Major Adverse Cardiovascular Events (MACE)
Description: MACE was defined as all-cause death, adjudicated myocardial infarction, stroke/transient ischemic attack, heart failure or recurrent ischemia requiring urgent revascularization.
Time Frame: Up to Week 14
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 135 | 199 | 192 | 391
Participants | 23 | 28 | 34 | 62
Statistical Analysis 1: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Test type: Superiority; p = 0.4110, Cox' proportional hazards model; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.46 to 1.38]
Statistical Analysis 2: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Test type: Superiority; p = 0.9318, Cox' proportional hazards model; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.60 to 1.74]
Statistical Analysis 3: Comparison: Placebo (P) vs A and B Combined (C); Test type: Superiority; p = 0.6805, Cox' proportional hazards model; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.56 to 1.46]

3. Primary Outcome: Number of Participants With Any Pure MACE
Description: Pure MACE was defined as all-cause death, adjudicated myocardial infarction or stroke/transient ischemic attack.
Time Frame: Up to Week 14
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 135 | 199 | 192 | 391
Participants | 19 | 21 | 29 | 50
Statistical Analysis 1: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Test type: Superiority or Other; p = 0.2990, Cox' proportional hazards model; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.39 to 1.34]
Statistical Analysis 2: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Test type: Superiority or Other; p = 0.8235, Cox' proportional hazards model; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.60 to 1.90]
Statistical Analysis 3: Comparison: Placebo (P) vs A and B Combined (C); Test type: Superiority or Other; p = 0.6590, Cox' proportional hazards model; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.52 to 1.51]

4. Primary Outcome: Number of Participants With Hematology Data of Potential Clinical Importance (PCI) at Any Visit Post-Baseline
Description: Hematology parameters (PCI range): Eosinophils (<0.045 or >0.605 Giga cells per liter [GI/L]), Hematocrit (<0.297 or >0.506 ratio), Hemoglobin (<85 or >200 grams per liter [g/L]), Lymphocytes (<0.765 or >4.51GI/L), Mean Corpuscle Hemoglobin (MCH) (<24.3 or >38.5 picograms [PG]), Mean Corpuscle Hemoglobin Concentration (MCHC) (<256 or >432 g/L), Mean Corpuscle Volume (MCV) (<70 or >115 femtoliter [FL]), Monocytes (<0.18 or >1.21 GI/L), Platelet count (<104 or >480 GI/L), Red Cell Distribution Width (RDW) (<7.2 or >18%), Red Blood Cell (RBC) count (<2.88 or >6.12 trillion per liter [TI/L] for females and <3.52 or >6.96 TI/L for males) , Reticulocytes (<22.5 or >93.5 10^9/L), Total Absolute Neutrophil Count (ANC) (<1.62 or >8.8 GI/L), White Blood Cell (WBC) count (<3.04 or >12 GI/L) were analyzed. The data was presented as High and low, at any visit post-Baseline. Only parameters with observed abnormal values were presented.
Time Frame: Up to Week 14
Population: Safety Population. Number of participants with analyzable samples at the time of analysis were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 120 | 173 | 166 | 339
Participants
  Eosinophils, high | 2 | 7 | 11 | 18
  Eosinophils, low | 14 | 20 | 16 | 36
  Hematocrit, high | 2 | 5 | 5 | 10
  Hematocrit, low | 2 | 8 | 8 | 16
  Hemoglobin, high | 0 | 1 | 0 | 1
  Hemoglobin, low | 0 | 1 | 2 | 3
  Lymphocytes, high | 0 | 1 | 2 | 3
  Lymphocytes, low | 2 | 7 | 5 | 12
  MCH, low | 0 | 1 | 2 | 3
  Monocytes, high | 1 | 1 | 3 | 4
  Monocytes, low | 14 | 15 | 19 | 34
  Platelet count, high | 0 | 4 | 3 | 7
  Platelet count, low | 2 | 1 | 2 | 3
  RDW, high | 3 | 3 | 7 | 10
  RBC count, high | 0 | 1 | 0 | 1
  RBC count, low | 10 | 10 | 11 | 21
  Reticulocytes, high | 30 | 49 | 36 | 85
  Reticulocytes, low | 5 | 4 | 4 | 8
  ANC, high | 4 | 12 | 19 | 31
  ANC, low | 1 | 2 | 0 | 2
  WBC count, high | 5 | 11 | 15 | 26

5. Primary Outcome: Number of Participants With Clinical Chemistry Data of PCI at Any Visit Post-Baseline
Description: Clinical chemistry parameters (PCI range): Alanine Amino Transferase (ALT) (>=3x upper limit normal [ULN] units per liter [U/L]), Albumin (<25.6 or >60 g/L), Alkaline Phosphatase (>=2x ULN U/L), Aspartate Amino Transferase (AST) (>=3x ULN U/L), Calcium (<2.0776 or >2.6112 millimoles per liter [mmol/L]), Carbon dioxide content/Bicarbonate (CO2/HCO3) (<19.6 or >32.64 mmol/L), Chloride (<93.1 or >110.16 mmol/L), Creatinine (<39.6 or >136.4 micromole per liter [µmol/L]) , Glucose (<3.51 or >6.05 mmol/L), Potassium (<3.43 or >5.406 mmol/L), Sodium (<132.3 or >148.92 mmol/L), Total Bilirubin (T. bilirubin) (>=1.5xULN µmol/L) , Total Protein (<50 or >95 g/L), Urea/Blood urea nitrogen (BUN) (<2.25 or >11.55 mmol/L) and Uric acid (<135 or >495 µmol/L) were analyzed. The data was presented as High and low, at any visit post-Baseline. Only parameters with observed abnormal values were presented.
Time Frame: Up to Week 14
Population: Safety Population. Number of participants with analyzable samples at the time of analysis were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 135 | 199 | 192 | 391
Participants
  ALT, high: number analyzed (Participants) | 124 | 177 | 173 | 350
  ALT, high | 1 | 4 | 2 | 6
  Albumin, low: number analyzed (Participants) | 122 | 175 | 170 | 345
  Albumin, low | 0 | 0 | 1 | 1
  Alkaline phosphatase, high: number analyzed (Participants) | 127 | 183 | 185 | 368
  Alkaline phosphatase, high | 0 | 2 | 0 | 2
  AST, high: number analyzed (Participants) | 124 | 177 | 173 | 350
  AST, high | 0 | 2 | 2 | 4
  Calcium, high: number analyzed (Participants) | 121 | 175 | 170 | 345
  Calcium, high | 4 | 3 | 5 | 8
  Calcium, low: number analyzed (Participants) | 121 | 175 | 170 | 345
  Calcium, low | 9 | 17 | 15 | 32
  CO2/HCO3, high: number analyzed (Participants) | 121 | 175 | 170 | 345
  CO2/HCO3, high | 1 | 1 | 3 | 4
  CO2/HCO3, low: number analyzed (Participants) | 121 | 175 | 170 | 345
  CO2/HCO3, low | 39 | 61 | 76 | 137
  Chloride, high: number analyzed (Participants) | 122 | 175 | 170 | 345
  Chloride, high | 1 | 5 | 6 | 11
  Chloride, low: number analyzed (Participants) | 122 | 175 | 170 | 345
  Chloride, low | 0 | 3 | 1 | 4
  Creatinine, high: number analyzed (Participants) | 122 | 175 | 170 | 345
  Creatinine, high | 6 | 10 | 17 | 27
  Creatinine, low: number analyzed (Participants) | 122 | 175 | 170 | 345
  Creatinine, low | 0 | 1 | 0 | 1
  Glucose, high: number analyzed (Participants) | 122 | 175 | 169 | 344
  Glucose, high | 90 | 132 | 113 | 245
  Glucose, low: number analyzed (Participants) | 122 | 175 | 169 | 344
  Glucose, low | 3 | 0 | 2 | 2
  Potassium, high: number analyzed (Participants) | 120 | 175 | 170 | 345
  Potassium, high | 0 | 6 | 4 | 10
  Potassium, low: number analyzed (Participants) | 120 | 175 | 170 | 345
  Potassium, low | 3 | 1 | 4 | 5
  Sodium, high: number analyzed (Participants) | 122 | 175 | 169 | 344
  Sodium, high | 0 | 1 | 1 | 2
  Sodium, low: number analyzed (Participants) | 122 | 175 | 169 | 344
  Sodium, low | 1 | 6 | 2 | 8
  T. Bilirubin, high: number analyzed (Participants) | 124 | 177 | 173 | 350
  T. Bilirubin, high | 0 | 3 | 0 | 3
  Total protein, low: number analyzed (Participants) | 122 | 175 | 170 | 345
  Total protein, low | 0 | 2 | 3 | 5
  Urea/BUN, high: number analyzed (Participants) | 122 | 175 | 170 | 345
  Urea/BUN, high | 4 | 8 | 15 | 23
  Urea/BUN, low: number analyzed (Participants) | 122 | 175 | 170 | 345
  Urea/BUN, low | 0 | 0 | 1 | 1
  Uric acid, high: number analyzed (Participants) | 122 | 175 | 170 | 345
  Uric acid, high | 19 | 29 | 29 | 58
  Uric acid, low: number analyzed (Participants) | 122 | 175 | 170 | 345
  Uric acid, low | 0 | 1 | 0 | 1

6. Primary Outcome: Number of Participants With Liver Function Test Elevations at Any Time Post-Baseline
Description: Liver function test parameters: Alanine aminotransferase (ALT), Total Bilirubin (T. Bilirubin), Aspartate aminotransferase (AST), Alkaline Phosphatase, Gamma glutamyl transferase (GGT) and Creatine Kinase were analyzed and presented as elevated test values at any time post-Baseline. The elevations were presented as >=2xULN, >=3xULN, >=5xULN, >=10xULN, and >=20xULN. n= number of participants with at least one non-missing result of the particular lab test post-Baseline.
Time Frame: Up to Week 14
Population: Safety Population. Number of participants with analyzable samples at the time of analysis were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 135 | 199 | 192 | 391
Participants
  ALT, >=2xULN: number analyzed (Participants) | 124 | 177 | 173 | 350
  ALT, >=2xULN | 4 | 7 | 4 | 11
  ALT, >=3xULN: number analyzed (Participants) | 124 | 177 | 173 | 350
  ALT, >=3xULN | 1 | 4 | 2 | 6
  ALT, >=5xULN: number analyzed (Participants) | 124 | 177 | 173 | 350
  ALT, >=5xULN | 0 | 3 | 0 | 3
  T. Bilirubin, >=1.5xULN: number analyzed (Participants) | 124 | 177 | 173 | 350
  T. Bilirubin, >=1.5xULN | 0 | 3 | 0 | 3
  AST, >=2xULN: number analyzed (Participants) | 124 | 177 | 173 | 350
  AST, >=2xULN | 3 | 10 | 3 | 13
  AST, >=3xULN: number analyzed (Participants) | 124 | 177 | 173 | 350
  AST, >=3xULN | 0 | 2 | 2 | 4
  AST, >=5xULN: number analyzed (Participants) | 124 | 177 | 173 | 350
  AST, >=5xULN | 0 | 1 | 0 | 1
  Alkaline phosphatase, >=1.5xULN: number analyzed (Participants) | 122 | 176 | 170 | 346
  Alkaline phosphatase, >=1.5xULN | 0 | 3 | 2 | 5
  Alkaline phosphatase, >=2xULN: number analyzed (Participants) | 122 | 176 | 170 | 346
  Alkaline phosphatase, >=2xULN | 0 | 2 | 1 | 3
  Alkaline phosphatase, >=3xULN: number analyzed (Participants) | 122 | 176 | 170 | 346
  Alkaline phosphatase, >=3xULN | 0 | 1 | 0 | 1
  Alkaline phosphatase, >=5xULN: number analyzed (Participants) | 122 | 176 | 170 | 346
  Alkaline phosphatase, >=5xULN | 0 | 1 | 0 | 1
  GGT, >=2xULN: number analyzed (Participants) | 122 | 175 | 170 | 345
  GGT, >=2xULN | 11 | 13 | 12 | 25
  GGT, >=3xULN: number analyzed (Participants) | 122 | 175 | 170 | 345
  GGT, >=3xULN | 5 | 5 | 4 | 9
  GGT, >=5xULN: number analyzed (Participants) | 122 | 175 | 170 | 345
  GGT, >=5xULN | 1 | 2 | 2 | 4
  Creatine kinase, >=2xULN: number analyzed (Participants) | 1 | 5 | 3 | 8
  Creatine kinase, >=2xULN | 0 | 1 | 0 | 1

7. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings at Any Time Post-Baseline
Description: A single 12-lead ECG was obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT corrected (QTc) intervals. ECG findings were presented as Normal, Abnormal - Not clinically significant and Abnormal - Clinically significant at any time post-Baseline.
Time Frame: Up to Week 14
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 125 | 182 | 180 | 362
Participants
  Normal | 34 | 41 | 40 | 81
  Abnormal - Not clinically significant | 77 | 115 | 118 | 233
  Abnormal - clinically significant | 14 | 26 | 22 | 48

8. Primary Outcome: Number of Participants With Vital Signs of PCI at Any Visit Post-Baseline
Description: Vital signs (PCI range): Systolic blood pressure (SBP) (<75 and >200 millimeter of mercury [mmHg]), Diastolic blood pressure (DBP) (<40 and >120 mmHg) and Heart rate (<30 and >200 beats per minute [bpm]) were analyzed and were presented at any visit post-Baseline. Participants with both Normal and Low values were counted once under their worst case (Low). Participants with both Normal and High values were counted once under their worst case (High). Participants with both High and Low values were counted under both categories. All heart rate values were within normal range, hence not presented.
Time Frame: Up to Week 14
Population: Safety Population. Number of participants with analyzable samples at the time of analysis were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 132 | 192 | 189 | 381
Participants
  DBP, high | 0 | 0 | 2 | 2
  DBP, low | 1 | 1 | 1 | 2
  SBP, high | 0 | 1 | 0 | 1
  SBP, low | 0 | 1 | 0 | 1

9. Primary Outcome: Mean High-sensitive C-Reactive Protein (hsCRP) Value at Week 12
Description: Analysis of hsCRP included all participants who provided data at Baseline and at least one post-Baseline measure. Statistical analyses was performed to compare hsCRP levels between study drug and placebo. Log transformed ratio to Baseline hsCRP was analyzed using repeated measures analysis of covariance (ANCOVA) including a term for treatment, adjusting for Baseline hsCRP as a covariate, and accounting for other covariates as appropriate to the study design.
Time Frame: At Week 12
Population: Intent-to-treat (ITT) Population comprised all randomized participants who received at least one dose of study medication and at least one on treatment assessment. Only those participants with data available at Week 12 were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg per liter (mg/L)
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 87 | 105 | 109 | 214
mg per liter (mg/L) | 1.52 (153.7) | 1.30 (183.5) | 1.46 (164.4) | 1.38 (173.3)
Statistical Analysis 1: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Test type: Superiority; p = 0.151, Repeated measures ANCOVA; test to reference ratio = 0.80, 95% CI 2-sided [0.59 to 1.09]
Statistical Analysis 2: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Test type: Superiority; p = 0.744, Repeated measures ANCOVA; test to reference ratio = 0.95, 95% CI 2-sided [0.70 to 1.29]
Statistical Analysis 3: Comparison: Placebo (P) vs A and B Combined (C); Test type: Superiority; p = 0.317, Repeated measures ANCOVA; test to treatment ratio = 0.87, 95% CI 2-sided [0.66 to 1.14]

10. Primary Outcome: Mean Cardiac Troponin I (cTnI) Area Under Concentration-time Curve (AUC) Over 72 Hours Post-randomization or Until Hospital Discharge (Whichever Comes First)
Description: cTnI AUC was the average concentration of cTnI during hospital stay. Statistical analyses was performed to compare cTnI levels between study drug and placebo, via ANCOVA.
Time Frame: At pre-dose and at 8, 16, 24, 32, 40, 48, 56, 64 and 72 hours
Population: ITT Population. Only those participants available at 72 hours were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nonograms*hour per milliliter (ng*hr/mL)
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 48 | 75 | 74 | 149
nonograms*hour per milliliter (ng*hr/mL) | 1.7 (469.3) | 1.1 (397.6) | 1.3 (586.6) | 1.2 (478.9)
Statistical Analysis 1: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Test type: Superiority; p = 0.83, ANCOVA; test to reference ratio = 1.03, 95% CI 2-sided [0.80 to 1.32]
Statistical Analysis 2: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Test type: Superiority; p = 0.56, ANCOVA; test to reference ratio = 1.08, 95% CI 2-sided [0.84 to 1.39]
Statistical Analysis 3: Comparison: Placebo (P) vs A and B Combined (C); Test type: Superiority; p = 0.65, ANCOVA; test to reference ratio = 1.05, 95% CI 2-sided [0.84 to 1.32]

11. Secondary Outcome: Mean hsCRP Over Hospitalization Period and Through Week 14
Description: Analysis of hsCRP included all participants who provided data at Baseline and at least one post-Baseline measure. The sample had a collection window of +/- 8 hours. Statistical analyses was performed to compare hsCRP levels between study drug and placebo. Log transformed ratio to Baseline hsCRP was analyzed using ANCOVA including a term for treatment, adjusting for Baseline hsCRP as a covariate, and accounting for other covariates as appropriate to the study design.
Time Frame: Up to Week 14
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 138 | 196 | 192 | 388
mg/L
  Predose: number analyzed (Participants) | 131 | 186 | 178 | 364
  Predose | 4.03 (232.4) | 4.26 (263.8) | 4.31 (210.1) | 4.29 (235.7)
  24 hours: number analyzed (Participants) | 104 | 148 | 139 | 287
  24 hours | 9.10 (241.8) | 6.76 (325.1) | 6.07 (259.9) | 6.41 (291.3)
  48 hours: number analyzed (Participants) | 73 | 104 | 98 | 202
  48 hours | 14.82 (236.8) | 7.53 (306.3) | 6.69 (335.6) | 7.11 (318.7)
  72 hours: number analyzed (Participants) | 52 | 77 | 76 | 153
  72 hours | 15.34 (300.8) | 7.92 (314.6) | 6.91 (337.6) | 7.40 (323.8)
  Discharge/Early withdrawal: number analyzed (Participants) | 89 | 127 | 123 | 250
  Discharge/Early withdrawal | 8.95 (171.3) | 6.46 (292.5) | 4.82 (214.5) | 5.59 (253.9)
  Week 2: number analyzed (Participants) | 96 | 128 | 130 | 258
  Week 2 | 3.30 (232.6) | 2.30 (302.9) | 2.18 (319.3) | 2.24 (309.6)
  Week 4: number analyzed (Participants) | 95 | 112 | 109 | 221
  Week 4 | 1.85 (203.0) | 1.42 (227.0) | 1.66 (214.8) | 1.54 (220.7)
  Week 8: number analyzed (Participants) | 90 | 109 | 109 | 218
  Week 8 | 1.65 (160.7) | 1.36 (198.0) | 1.50 (193.1) | 1.43 (195.0)
  Week 14: number analyzed (Participants) | 87 | 107 | 111 | 218
  Week 14 | 1.60 (172.5) | 2.47 (187.0) | 2.59 (168.9) | 2.53 (177.0)
Statistical Analysis 1: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Placebo (P) vs Losmapimod 7.5 mg (A): For 24 hours; Test type: Superiority; p = 0.040, Repeated measures ANCOVA; Test to reference ratio = 0.77, 95% CI 2-sided [0.60 to 0.99]
Statistical Analysis 2: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Placebo (P) vs Losmapimod 15 mg followed by Losmapimod 7.5 mg (B): For 24 hours; Test type: Superiority; p = 0.001, Repeated measures ANCOVA; test to reference ratio = 0.66, 95% CI 2-sided [0.52 to 0.85]
Statistical Analysis 3: Comparison: Placebo (P) vs A and B Combined (C); Placebo (P) vs A and B Combined (C): For 24 hours; Test type: Superiority; p = 0.003, Repeated measures ANCOVA; test to reference ratio = 0.71, 95% CI 2-sided [0.57 to 0.89]
Statistical Analysis 4: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Placebo (P) vs Losmapimod 7.5 mg (A): For 48 hours; Test type: Superiority; p < 0.001, Repeated measures ANCOVA; test to reference ratio = 0.56, 95% CI 2-sided [0.40 to 0.78]
Statistical Analysis 5: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Placebo (P) vs Losmapimod 15 mg followed by Losmapimod 7.5 mg (B): For 48 hours; Test type: Superiority; p < 0.001, Repeated measures ANCOVA; test to reference ratio = 0.47, 95% CI 2-sided [0.33 to 0.65]
Statistical Analysis 6: Comparison: Placebo (P) vs A and B Combined (C); Placebo (P) vs A and B Combined (C): For 48 hours; Test type: Superiority; p < 0.001, Repeated measures ANCOVA; test to reference ratio = 0.51, 95% CI 2-sided [0.38 to 0.69]
Statistical Analysis 7: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Placebo (P) vs Losmapimod 7.5 mg (A): For 72 hours; Test type: Superiority; p = 0.059, Repeated measures ANCOVA; test to reference ratio = 0.68, 95% CI 2-sided [0.45 to 1.01]
Statistical Analysis 8: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Placebo (P) vs Losmapimod 15 mg followed by Losmapimod 7.5 mg (B): For 72 hours; Test type: Superiority; p = 0.013, Repeated measures ANCOVA; test to reference ratio = 0.60, 95% CI 2-sided [0.40 to 0.90]
Statistical Analysis 9: Comparison: Placebo (P) vs A and B Combined (C); Placebo (P) vs A and B Combined (C): For 72 hours; Test type: Superiority; p = 0.015, Repeated measures ANCOVA; test to reference ratio = 0.64, 95% CI 2-sided [0.45 to 0.92]
Statistical Analysis 10: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Placebo (P) vs Losmapimod 7.5 mg (A): For Week 2; Test type: Superiority; p = 0.073, Repeated measures ANCOVA; test to reference ratio = 0.70, 95% CI 2-sided [0.48 to 1.03]
Statistical Analysis 11: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Placebo (P) vs Losmapimod 15 mg followed by Losmapimod 7.5 mg (B): For Week 2; Test type: Superiority; p = 0.075, Repeated measures ANCOVA; test to reference ratio = 0.70, 95% CI 2-sided [0.48 to 1.04]
Statistical Analysis 12: Comparison: Placebo (P) vs A and B Combined (C); Placebo (P) vs A and B Combined (C): For Week 2; Test type: Superiority; p = 0.044, Repeated measures ANCOVA; test to reference ratio = 0.70, 95% CI 2-sided [0.50 to 0.99]
Statistical Analysis 13: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Placebo (P) vs Losmapimod 7.5 mg (A): For Week 4; Test type: Superiority; p = 0.157, Repeated measures ANCOVA; test to reference ratio = 0.78, 95% CI 2-sided [0.55 to 1.10]
Statistical Analysis 14: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Placebo (P) vs Losmapimod 15 mg followed by Losmapimod 7.5 mg (B): For Week 4; Test type: Superiority; p = 0.548, ANCOVA; test to reference ratio = 0.90, 95% CI 2-sided [0.63 to 1.28]
Statistical Analysis 15: Comparison: Placebo (P) vs A and B Combined (C); Placebo (P) vs A and B Combined (C): For Week 4; Test type: Superiority; p = 0.253, Repeated measures ANCOVA; test to reference ratio = 0.83, 95% CI 2-sided [0.61 to 1.14]
Statistical Analysis 16: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Placebo (P) vs Losmapimod 7.5 mg (A): For Week 8; Test type: Superiority; p = 0.204, Repeated measures ANCOVA; test to reference ratio = 0.80, 95% CI 2-sided [0.58 to 1.13]
Statistical Analysis 17: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Placebo (P) vs Losmapimod 15 mg followed by Losmapimod 7.5 mg (B): For Week 8; Test type: Superiority; p = 0.965, Repeated measures ANCOVA; test to reference ratio = 0.99, 95% CI 2-sided [0.71 to 1.39]
Statistical Analysis 18: Comparison: Placebo (P) vs A and B Combined (C); Placebo (P) vs A and B Combined (C): For Week 8; Test type: Superiority; p = 0.457, Repeated measures ANCOVA; test to reference ratio = 0.89, 95% CI 2-sided [0.66 to 1.20]
Statistical Analysis 19: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Placebo (P) vs Losmapimod 7.5 mg (A): For Week 14; Test type: Superiority; p = 0.008, Repeated measures ANCOVA; test to reference ratio = 1.58, 95% CI 2-sided [1.13 to 2.22]
Statistical Analysis 20: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Placebo (P) vs Losmapimod 15 mg followed by Losmapimod 7.5 mg (B): For Week 14; Test type: Superiority; p = 0.002, Repeated measures ANCOVA; test to reference ratio = 1.69, 95% CI 2-sided [1.21 to 2.38]
Statistical Analysis 21: Comparison: Placebo (P) vs A and B Combined (C); Placebo (P) vs A and B Combined (C): For Week 14; Test type: Superiority; p = 0.001, Repeated measures ANCOVA; test to reference ratio = 1.64, 95% CI 2-sided [1.21 to 2.21]

12. Secondary Outcome: Mean Interleukin-6 (IL-6) Value at 24 Hours Post-randomization and at Weeks 2 and 12
Description: Statistical analyses was performed to compare IL-6 levels between study drug and placebo. Log transformed ratio to Baseline IL-6 was analyzed using repeated measures ANCOVA including a term for treatment, adjusting for Baseline IL-6 as a covariate, and accounting for other covariates as appropriate to the study design.
Time Frame: 24 hours post-randomization and at Weeks 2 and 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms per milliliter (pg/mL)
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 138 | 196 | 192 | 388
picograms per milliliter (pg/mL)
  24 hours: number analyzed (Participants) | 102 | 147 | 142 | 289
  24 hours | 10.59 (147.8) | 6.08 (144.6) | 7.11 (148.6) | 6.57 (146.8)
  Week 2: number analyzed (Participants) | 101 | 134 | 134 | 268
  Week 2 | 3.50 (140.6) | 2.75 (116.1) | 3.14 (111.6) | 2.94 (114.0)
  Week 12: number analyzed (Participants) | 93 | 110 | 113 | 223
  Week 12 | 2.62 (102.8) | 2.29 (96.0) | 2.61 (88.4) | 2.45 (92.3)
Statistical Analysis 1: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Placebo (P) vs Losmapimod 7.5 mg (A): For 24 hours; Test type: Superiority; p < 0.001, Repeated measures ANCOVA; test to reference ratio = 0.54, 95% CI 2-sided [0.43 to 0.69]
Statistical Analysis 2: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Placebo (P) vs Losmapimod 15 mg followed by Losmapimod 7.5 mg (B): For 24 hours; Test type: Superiority; p < 0.001, Repeated measures ANCOVA; test to reference ratio = 0.64, 95% CI 2-sided [0.50 to 0.82]
Statistical Analysis 3: Comparison: Placebo (P) vs A and B Combined (C); Placebo (P) vs A and B Combined (C): For 24 hours; Test type: Superiority; p < 0.001, Repeated measures ANCOVA; test to reference ratio = 0.59, 95% CI 2-sided [0.48 to 0.73]
Statistical Analysis 4: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Placebo (P) vs Losmapimod 7.5 mg (A): For Week 2; Test type: Superiority; p = 0.031, Repeated measures ANCOVA; test to reference ratio = 0.76, 95% CI 2-sided [0.59 to 0.98]
Statistical Analysis 5: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Placebo (P) vs Losmapimod 15 mg followed by Losmapimod 7.5 mg (B): For Week 2; Test type: Superiority; p = 0.315, Repeated measures ANCOVA; test to reference ratio = 0.88, 95% CI 2-sided [0.68 to 1.13]
Statistical Analysis 6: Comparison: Placebo (P) vs A and B Combined (C); Placebo (P) vs A and B Combined (C): For Week 2; Test type: Superiority; p = 0.075, Repeated measures ANCOVA; test to reference ratio = 0.82, 95% CI 2-sided [0.65 to 1.02]
Statistical Analysis 7: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Placebo (P) vs Losmapimod 7.5 mg (A): For Week 12; Test type: Superiority; p = 0.068, Repeated measures ANCOVA; test to reference ratio = 0.81, 95% CI 2-sided [0.65 to 1.02]
Statistical Analysis 8: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Placebo (P) vs Losmapimod 15 mg followed by Losmapimod 7.5 mg (B): For Week 12; Test type: Superiority; p = 0.824, Repeated measures ANCOVA; test to reference ratio = 0.97, 95% CI 2-sided [0.78 to 1.22]
Statistical Analysis 9: Comparison: Placebo (P) vs A and B Combined (C); Placebo (P) vs A and B Combined (C): For Week 12; Test type: Superiority; p = 0.246, Repeated measures ANCOVA; test to reference ratio = 0.89, 95% CI 2-sided [0.73 to 1.09]

13. Secondary Outcome: Mean Creatine Kinase (MB Isoenzyme) (CK-MB) AUC Over 72 Hours Post-randomization or Until Hospital Discharge (Whichever Comes First)
Description: Statistical analyses was performed to compare CK-MB levels between study drug and placebo. Log transformed ratio to Baseline CK-MB was analyzed using repeated measures ANCOVA including a term for treatment, adjusting for Baseline CK-MB as a covariate, and accounting for other covariates as appropriate to the study design.
Time Frame: At pre-dose and at hours 8, 16, 24, 32, 40, 48, 56, 64 and 72
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 138 | 196 | 192 | 388
ng*hr/mL
  Predose: number analyzed (Participants) | 128 | 176 | 167 | 343
  Predose | 11.5 (247.9) | 10.5 (196.4) | 9.8 (233.5) | 10.2 (213.5)
  8 hours: number analyzed (Participants) | 107 | 172 | 155 | 327
  8 hours | 9.0 (234.5) | 7.8 (185.0) | 8.4 (242.2) | 8.1 (210.4)
  16 hours: number analyzed (Participants) | 105 | 162 | 151 | 313
  16 hours | 7.1 (194.2) | 6.5 (170.9) | 7.0 (213.7) | 6.8 (190.4)
  24 hours: number analyzed (Participants) | 97 | 138 | 134 | 272
  24 hours | 6.2 (151.1) | 5.2 (147.2) | 6.1 (171.8) | 5.6 (159.3)
  32 hours: number analyzed (Participants) | 84 | 127 | 124 | 251
  32 hours | 4.1 (139.5) | 4.5 (129.5) | 5.1 (130.4) | 4.8 (129.9)
  40 hours: number analyzed (Participants) | 78 | 117 | 113 | 230
  40 hours | 3.2 (119.3) | 3.6 (110.1) | 4.0 (118.9) | 3.8 (114.3)
  48 hours: number analyzed (Participants) | 63 | 96 | 92 | 188
  48 hours | 3.0 (103.1) | 3.2 (110.0) | 3.3 (103.3) | 3.3 (106.3)
  56 hours: number analyzed (Participants) | 52 | 84 | 72 | 156
  56 hours | 2.5 (81.5) | 2.8 (98.3) | 3.1 (91.9) | 2.9 (95.2)
  64 hours: number analyzed (Participants) | 46 | 81 | 71 | 152
  64 hours | 2.2 (75.5) | 2.6 (97.8) | 3.0 (87.5) | 2.8 (93.0)
  72 hours: number analyzed (Participants) | 46 | 70 | 70 | 140
  72 hours | 2.4 (117.7) | 2.6 (94.3) | 2.8 (84.3) | 2.7 (89.1)
  DIS/EW: number analyzed (Participants) | 75 | 119 | 112 | 231
  DIS/EW | 2.9 (117.4) | 2.6 (96.4) | 2.9 (105.6) | 2.8 (100.8)
Statistical Analysis 1: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Placebo (P) vs Losmapimod 7.5 mg (A): For 72 hours; Test type: Superiority; p = 0.66, Repeated measures ANCOVA; test to reference ratio = 1.04, 95% CI 2-sided [0.89 to 1.21]
Statistical Analysis 2: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Placebo (P) vs Losmapimod 15 mg followed by Losmapimod 7.5 mg (B): For 72 hours; Test type: Superiority; p = 0.39, Repeated measures ANCOVA; test to reference ratio = 1.07, 95% CI 2-sided [0.92 to 1.25]
Statistical Analysis 3: Comparison: Placebo (P) vs A and B Combined (C); Placebo (P) vs A and B Combined (C): For 72 hours; Test type: Superiority; p = 0.47, Repeated measures ANCOVA; test to reference ratio = 1.05, 95% CI 2-sided [0.92 to 1.21]

14. Secondary Outcome: Peak cTnI Over 72 Hours Post-randomization or Until Hospital Discharge (Whichever Comes First)
Description: Statistical analyses was performed to compare cTnI levels between study drug and placebo. Log transformed ratio to Baseline cTnI was analyzed using repeated measures ANCOVA including a term for treatment, adjusting for Baseline cTnI as a covariate, and accounting for other covariates as appropriate to the study design.
Time Frame: Up to 72 hours
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 129 | 187 | 181 | 368
ng/mL | 4.02 (482.0) | 3.49 (575.3) | 3.54 (867.8) | 3.52 (701.0)
Statistical Analysis 1: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Test type: Superiority; p = 0.92, Repeated measures ANCOVA; test to reference ratio = 0.99, 95% CI 2-sided [0.78 to 1.25]
Statistical Analysis 2: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Test type: Superiority; p = 0.52, Repeated measures ANCOVA; test to reference ratio = 1.08, 95% CI 2-sided [0.85 to 1.36]
Statistical Analysis 3: Comparison: Placebo (P) vs A and B Combined (C); Test type: Superiority; p = 0.76, Repeated measures ANCOVA; test to reference ratio = 1.03, 95% CI 2-sided [0.84 to 1.27]

15. Secondary Outcome: Mean Brain Natriuretic Peptide (BNP) at Discharge and Week 12
Description: Statistical analyses was performed to compare BNP levels between study drug and placebo. Log transformed ratio to Baseline BNP was analyzed using repeated measures ANCOVA including a term for treatment, adjusting for Baseline BNP as a covariate, and accounting for other covariates as appropriate to the study design.
Time Frame: At discharge and Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 138 | 196 | 192 | 388
pg/mL
  Discharge/Early withdrawal: number analyzed (Participants) | 83 | 122 | 125 | 247
  Discharge/Early withdrawal | 72.56 (208.2) | 65.84 (174.8) | 73.24 (193.9) | 69.49 (183.9)
  Week 12: number analyzed (Participants) | 89 | 112 | 112 | 224
  Week 12 | 49.41 (167.1) | 37.41 (141.8) | 37.02 (159.8) | 37.22 (150.1)
Statistical Analysis 1: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Placebo (P) vs Losmapimod 7.5 mg (A): For discharge/early withdrawal; Test type: Superiority; p = 0.57, Repeated measures ANCOVA; test to reference ratio = 0.93, 95% CI 2-sided [0.72 to 1.20]
Statistical Analysis 2: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Placebo (P) vs Losmapimod 15 mg followed by Losmapimod 7.5 mg (B): For discharge/early withdrawal; Test type: Superiority; p = 0.52, Repeated measures ANCOVA; test to reference ratio = 0.92, 95% CI 2-sided [0.72 to 1.18]
Statistical Analysis 3: Comparison: Placebo (P) vs A and B Combined (C); Placebo (P) vs A and B Combined (C): For discharge/early withdrawal; Test type: Superiority; p = 0.50, Repeated measures ANCOVA; test to reference ratio = 0.92, 95% CI 2-sided [0.74 to 1.16]
Statistical Analysis 4: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Placebo (P) vs Losmapimod 7.5 mg (A): For Week 12; Test type: Superiority; p = 0.03, Repeated measures ANCOVA; test to reference ratio = 0.73, 95% CI 2-sided [0.55 to 0.96]
Statistical Analysis 5: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Placebo (P) vs Losmapimod 15 mg followed by Losmapimod 7.5 mg (B): For Week 12; Test type: Superiority; p = 0.14, Repeated measures ANCOVA; test to reference ratio = 0.81, 95% CI 2-sided [0.61 to 1.07]
Statistical Analysis 6: Comparison: Placebo (P) vs A and B Combined (C); Placebo (P) vs A and B Combined (C): For Week 12; Test type: Superiority; p = 0.04, Repeated measures ANCOVA; test to reference ratio = 0.76, 95% CI 2-sided [0.60 to 0.98]

16. Secondary Outcome: Mean Infarct Size Prior to Discharge From Hospital (Approximately Day 3) and at Week 12
Description: Statistical analyses was performed to compare the infarct size (via MRI) at Week 12 via repeated measures ANOVA between study drug and placebo using Bayesian methods for inference. Myocardial infarct size was measured by delayed enhancement magnetic resonance imaging (MRI) as: Infarct size (% of left ventricular myocardium [% of LV]) for infarct 1. The infarct region 1 was the infarct region which the MRI interpretation process identified as the primary infarct region of the index hospitalization. Participants were included in the analyses, provided they have data for derivation of the measures of interest (MR infarct size). A total of 15 participants out of 93 MRI ITT participants were excluded from the analysis due to missing Baseline cTnI (10 participants) and onset chest pain duration (9 participants). Four participants had both covariate values missing.
Time Frame: Prior to discharge (visit 1) and at Week 12
Population: MRI ITT Population was subset of participants in the ITT Population who had at least one MRI scan. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent of left ventricle
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 26 | 37 | 30 | 67
Percent of left ventricle
  Day 3-5 (Visit 1): number analyzed (Participants) | 24 | 36 | 29 | 65
  Day 3-5 (Visit 1) | 7.804 (7.4066) | 5.575 (6.0525) | 5.848 (7.6326) | 5.697 (6.7483)
  Week 12: number analyzed (Participants) | 20 | 24 | 26 | 50
  Week 12 | 5.620 (5.4493) | 4.783 (5.2992) | 4.335 (5.9772) | 4.550 (5.6090)
Statistical Analysis 1: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Placebo (P) vs Losmapimod 7.5 mg (A): For Day 3-5 (visit 1); Test type: Superiority; p = 0.254, Repeated measures ANCOVA; Mean Difference (Final Values) = -1.92, 95% CI 2-sided [-5.25 to 1.41]
Statistical Analysis 2: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Placebo (P) vs Losmapimod 15 mg followed by Losmapimod 7.5 mg (B): For Day 3-5 (visit 1); Test type: Superiority; p = 0.106, Repeated measures ANCOVA; Mean Difference (Final Values) = -2.84, 95% CI 2-sided [-6.29 to 0.62]
Statistical Analysis 3: Comparison: Placebo (P) vs A and B Combined (C); Placebo (P) vs A and B Combined (C): For Day 3-5 (visit 1); Test type: Superiority; p = 0.126, Repeated measures ANCOVA; Mean Difference (Final Values) = -2.38, 95% CI 2-sided [-5.44 to 0.69]
Statistical Analysis 4: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Placebo (P) vs Losmapimod 7.5 mg (A): For Week 12; Test type: Superiority; p = 0.184, Repeated measures ANCOVA; Mean Difference (Final Values) = -1.91, 95% CI 2-sided [-4.74 to 0.92]
Statistical Analysis 5: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Placebo (P) vs Losmapimod 15 mg followed by Losmapimod 7.5 mg (B): For Week 12; Test type: Superiority; p = 0.093, Repeated measures ANCOVA; Mean Difference (Final Values) = -2.47, 95% CI 2-sided [-5.37 to 0.43]
Statistical Analysis 6: Comparison: Placebo (P) vs A and B Combined (C); Placebo (P) vs A and B Combined (C): For Week 12; Test type: Superiority; p = 0.096, Repeated measures ANCOVA; Mean Difference (Final Values) = -2.19, 95% CI 2-sided [-4.78 to 0.40]

17. Secondary Outcome: Mean Percent Left Ventricular Ejection Fraction (LVEF) at Week 12
Description: Statistical analyses of the treatment differences was performed to compare the LVEF (via MRI) at Week 12, and for the change from Day 3 to Week 12 via repeated measures ANCOVA between study drug and placebo. Cardiac MRIs were performed at qualified sites on participants who agree to participate in the MRI sub-study. A total of 15 participants out of 93 MRI ITT participants were excluded from the analysis due to missing Baseline cTnI (10 participants) and onset chest pain duration (9 participants). Four participants had both covariate values missing.
Time Frame: At Week 12
Population: MRI ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 20 | 24 | 26 | 50
Percent | 56.615 (11.1103) | 59.571 (7.2745) | 59.738 (9.5443) | 59.658 (8.4453)
Statistical Analysis 1: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Test type: Superiority; p = 0.124, Repeated measures ANCOVA; Mean Difference (Final Values) = 4.22, 95% CI 2-sided [-1.18 to 9.62]
Statistical Analysis 2: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Test type: Superiority; p = 0.029, Repeated measures ANCOVA; Mean Difference (Final Values) = 6.05, 95% CI 2-sided [0.63 to 11.47]
Statistical Analysis 3: Comparison: Placebo (P) vs A and B Combined (C); Test type: Superiority; p = 0.039, Repeated measures ANCOVA; Mean Difference (Final Values) = 5.14, 95% CI 2-sided [0.28 to 10.00]

18. Secondary Outcome: Mean Left Ventricular End-diastolic Volume (LVEDV) and Left Ventricular End-systolic Volume (LVESV) at Week 12
Description: Statistical analyses of the treatment differences was performed to compare the LVEDV and LVESV (via MRI) at Week 12, and for the change from Day 3 to Week 12 via repeated measures ANCOVA between study drug and placebo. Cardiac MRIs were performed at qualified sites on participants who agree to participate in the MRI sub-study. A total of 15 participants out of 93 MRI ITT participants were excluded from the analysis due to missing Baseline cTnI (10 participants) and onset chest pain duration (9 participants). Four participants had both covariate values missing.
Time Frame: At Week 12
Population: MRI ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 20 | 24 | 26 | 50
mL
  LVEDV | 132.895 (35.5648) | 125.942 (30.2434) | 130.642 (27.1760) | 128.386 (28.4914)
  LVESV | 58.660 (24.8018) | 52.115 (19.4760) | 53.710 (20.8387) | 52.944 (20.0063)
Statistical Analysis 1: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Placebo (P) vs Losmapimod 7.5 mg (A): For LVEDV; Test type: Superiority; p = 0.025, Repeated measures ANCOVA; Mean Difference (Final Values) = -21.53, 95% CI 2-sided [-40.27 to -2.79]
Statistical Analysis 2: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Placebo (P) vs Losmapimod 15 mg followed by Losmapimod 7.5 mg (B): For LVEDV; Test type: Superiority; p = 0.053, Repeated measures ANCOVA; Mean Difference (Final Values) = -18.65, 95% CI 2-sided [-37.58 to 0.29]
Statistical Analysis 3: Comparison: Placebo (P) vs A and B Combined (C); Placebo (P) vs A and B Combined (C): For LVEDV; Test type: Superiority; p = 0.021, Repeated measures ANCOVA; Mean Difference (Final Values) = -20.09, 95% CI 2-sided [-37.01 to -3.18]
Statistical Analysis 4: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Placebo (P) vs Losmapimod 7.5 mg (A): For LVESV; Test type: Superiority; p = 0.024, Repeated measures ANCOVA; Mean Difference (Final Values) = -15.82, 95% CI 2-sided [-29.51 to -2.14]
Statistical Analysis 5: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Placebo (P) vs Losmapimod 15 mg followed by Losmapimod 7.5 mg (B): For LVESV; Test type: Superiority; p = 0.016, Repeated measures ANCOVA; Mean Difference (Final Values) = -17.22, 95% CI 2-sided [-31.14 to -3.29]
Statistical Analysis 6: Comparison: Placebo (P) vs A and B Combined (C); Placebo (P) vs A and B Combined (C): For LVESV; Test type: Superiority; p = 0.010, Repeated measures ANCOVA; Mean Difference (Final Values) = -16.52, 95% CI 2-sided [-28.91 to -4.13]

19. Secondary Outcome: Mean Left Ventricular Mass at Week 12
Description: Statistical analyses of the treatment differences was performed to compare the left ventricular mass (via MRI) at Week 12, and for the change from Day 3 to Week 12 via repeated measures ANCOVA between study drug and placebo.Cardiac MRIs were performed at qualified sites on participants who agree to participate in the MRI sub-study. A total of 15 participants out of 93 MRI ITT participants were excluded from the analysis due to missing Baseline cTnI (10 participants) and onset chest pain duration (9 participants). Four participants had both covariate values missing.
Time Frame: At Week 12
Population: MRI ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: grams (gm)
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 20 | 24 | 26 | 50
grams (gm) | 145.463 (36.9074) | 141.449 (40.5956) | 154.194 (42.3668) | 148.076 (41.6018)
Statistical Analysis 1: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Test type: Superiority; p = 0.109, Repeated measures ANCOVA; Mean Difference (Final Values) = -22.21, 95% CI 2-sided [-49.51 to 5.09]
Statistical Analysis 2: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Test type: Superiority; p = 0.614, Repeated measures ANCOVA; Mean Difference (Final Values) = -7.13, 95% CI 2-sided [-35.22 to 20.96]
Statistical Analysis 3: Comparison: Placebo (P) vs A and B Combined (C); Test type: Superiority; p = 0.243, Repeated measures ANCOVA; Mean Difference (Final Values) = -14.67, 95% CI 2-sided [-39.52 to 10.18]

20. Secondary Outcome: Mean Regional Wall Motion Score Index at Week 12
Description: Wall motion score index is a semi-quantitative analysis of regional systolic function. Each segment is analyzed individually and scored on the basis of its motion and systolic thickening. This score is a 5-level score defines as: 1=normokinesis or hyperkinesis, 2=hypokinesi, 3=akinesis, 4=dyskinesis, 5=aneurysm. Wall motion score index is derived as a sum of all scores divided by the number of segments visualized. Larger score index indicates higher degree of abnormalities. Cardiac MRIs were performed at qualified sites on participants who agree to participate in the MRI sub-study. A total of 15 participants out of 93 MRI ITT participants were excluded from the analysis due to missing Baseline cTnI (10 participants) and onset chest pain duration (9 participants). Four participants had both covariate values missing.
Time Frame: At Week 12
Population: MRI ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 20 | 23 | 26 | 49
Scores on a scale | 0.306 (0.4096) | 0.179 (0.2704) | 0.186 (0.3326) | 0.182 (0.3019)
Statistical Analysis 1: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Test type: Superiority; p = 0.023, Repeated measures ANCOVA; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.44 to -0.03]
Statistical Analysis 2: Comparison: Placebo (P) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Test type: Superiority; p = 0.021, Repeated measures ANCOVA; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.45 to -0.04]
Statistical Analysis 3: Comparison: Placebo (P) vs A and B Combined (C); Test type: Superiority; p = 0.011, Repeated measures ANCOVA; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.42 to -0.06]

21. Secondary Outcome: Mean Hyperenhancement Score Index at Week 12
Description: The myocardium was divided into 17 segments. A score ranging from 0 to 4 was visually attributed to each of the 17 segments according to the transmural extent of the hyperenhancement: score 0=0%, 1=>0-25%, 2=>25-50%, 3=>50-75% and 4=>75-100%. All these 17 scores were summed. The resulting summed score ranged in theory from 0 to 68 and was thereafter expressed as a percentage of the maximum possible score of 68, with higher percentages indicating hyper-enhancement in a greater percentage of the tissue in a greater number of segments. Cardiac MRIs were performed at qualified sites on participants who agree to participate in the MRI sub-study. A total of 15 participants out of 93 MRI ITT participants were excluded from the analysis due to missing Baseline cTnI (10 participants) and onset chest pain duration (9 participants). Four participants had both covariate values missing. Statistical analysis was performed on LS mean value using repeated measures ANCOVA.
Time Frame: At week 12
Population: MRI ITT Population. Only those participants with data available at week 12 were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Combined (C)
Number analyzed (Participants) | 20 | 24 | 26 | 50
Scores on a scale | 0.350 (0.2648) | 0.282 (0.3117) | 0.249 (0.3096) | 0.265 (0.3079)
Statistical Analysis 1: Comparison: Placebo (P) vs Losmapimod 7.5 mg (A); Test type: Superiority; p = 0.137, Repeated measures ANCOVA; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.26 to 0.04]
Statistical Analysis 2: Comparison: Losmapimod 7.5 mg (A) vs Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B); Test type: Superiority; p = 0.036, Repeated measures ANCOVA; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.32 to -0.01]
Statistical Analysis 3: Comparison: Placebo (P) vs A and B Combined (C); Test type: Superiority; p = 0.047, Repeated measures ANCOVA; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.28 to -0.00]

ADVERSE EVENTS:
Time Frame: SAEs and nSAEs were collected from start of study medication up to Week 14.
Description: SAEs and nSAEs were reported for safety Population which consisted of all participants randomized to treatment, who had taken at least one dose of study medication.
Groups:
- A and B Comb (C): A combined data for eligible participants from arm A and arm B were presented.
Arm/Group | Placebo (P) | Losmapimod 7.5 mg (A) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) | A and B Comb (C)
All-Cause Mortality (participants affected / at risk) | 4/135 | 4/199 | 10/192 | 14/391
Serious Adverse Events (participants affected / at risk) | 32/135 | 51/199 | 43/192 | 94/391
Other Adverse Events (participants affected / at risk) | 52/135 | 55/199 | 49/192 | 104/391
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (P) (N=135) | Losmapimod 7.5 mg (A) (N=199) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) (N=192) | A and B Comb (C) (N=391)
Acute myocardial infarction (Cardiac disorders) | 2 | 4 | 6 | 10
Angina unstable (Cardiac disorders) | 3 | 4 | 5 | 9
Myocardial infarction (Cardiac disorders) | 7 | 4 | 1 | 5
Angina pectoris (Cardiac disorders) | 4 | 1 | 3 | 4
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 3 | 5
Cardiac failure (Cardiac disorders) | 0 | 2 | 4 | 6
Cardiogenic shock (Cardiac disorders) | 1 | 2 | 2 | 4
Arrhythmia (Cardiac disorders) | 1 | 0 | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 1 | 3
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 2 | 2
Ventricular fibrillation (Cardiac disorders) | 1 | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 1
Dressler's syndrome (Cardiac disorders) | 0 | 1 | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 0 | 1 | 1
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0 | 1
Ventricular asystole (Cardiac disorders) | 0 | 1 | 0 | 1
Ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 2 | 3
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 1
Chest pain (General disorders) | 3 | 4 | 4 | 8
Non-cardiac chest pain (General disorders) | 1 | 0 | 2 | 2
Thrombosis in device (General disorders) | 2 | 0 | 1 | 1
Multi-organ failure (General disorders) | 1 | 0 | 1 | 1
Death (General disorders) | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 3
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 3
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1 | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1 | 1
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 1 | 1
Subclavian artery stenosis (Vascular disorders) | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0 | 1
Labyrinthitis (Infections and infestations) | 1 | 0 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 3 | 0 | 3
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1
Delusion (Psychiatric disorders) | 0 | 0 | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (P) (N=135) | Losmapimod 7.5 mg (A) (N=199) | Losmapimod 15 mg Followed by Losmapimod 7.5 mg (B) (N=192) | A and B Comb (C) (N=391)
Headache (Nervous system disorders) | 11 | 15 | 13 | 28
Dizziness (Nervous system disorders) | 10 | 11 | 7 | 18
Chest pain (General disorders) | 7 | 13 | 9 | 22
Fatigue (General disorders) | 10 | 4 | 5 | 9
Nausea (Gastrointestinal disorders) | 8 | 7 | 4 | 11
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 6 | 10
Haematoma (Vascular disorders) | 8 | 11 | 6 | 17
Nasopharyngitis (Infections and infestations) | 7 | 1 | 9 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 4 | 9
Atrial fibrillation (Cardiac disorders) | 7 | 3 | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.